CLINICAL TRIAL: NCT05354206
Title: Neural Facilitation of Stimulation-assisted Movements in People With Spinal Cord Injury
Brief Title: Neural Facilitation of Movements in People With SCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in funding, transitioned to new grant and project
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ismael Seáñez, Assistant Professor of Biomedical Engineering and Neurosurgery, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202111151
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; spinal cord stimulation; rehabilitation; neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: After baseline evaluations of the effect of transcutaneous SCS on single pulse responses, motor function, and a familiarization phase on a body-machine interface, participants will be randomly assigned to one of two arms in the study.
  Arm 1: Participants will receive interventions A and B and transcranial magnetic stimulation is used to evaluate the excitability of the corticospinal tract.
  Arm 2: Participants will receive interventions A and B and a loud auditory stimuli is used to evaluate the excitability of the reticulospinal tract.
  Arms 1 and 2 will run in parallel. Participants will perform interventions A and B in a randomized cross-over design. In both interventions A and B, participants will use their legs to control a computer cursor as transcutaneous spinal cord stimulation is delivered. Intervention A, participants perform a range-of-motion task, while in intervention B, participants perform a precision-control task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of motor evoked potentials during non-invasive spinal cord stimulation and leg movements (Experimental): This arm will receive the transcranial magnetic stimulation to evaluate the excitability of the corticospinal tract first then the arm will receive the loud auditory stimuli to evaluate the excitability of the reticulospinal track second.
  Interventions: Other: Electrophysiology assessment - corticospinal tract; Other: Training with some stimulation
- Reaction time evaluation during non-invasive spinal cord stimulation and leg movements (Experimental): This arm will receive the loud auditory stimuli to evaluate the excitability of the reticulospinal tract first then the arm will receive the transcranial magnetic stimulation to excite the corticospinal tract second
  Interventions: Other: Electrophysiology assessment - reticulospinal tract; Other: Training with some stimulation

INTERVENTIONS:
Other: Electrophysiology assessment - corticospinal tract — Kinematics and cortical spinal motor excitability
  Arms: Evaluation of motor evoked potentials during non-invasive spinal cord stimulation and leg movements
Other: Electrophysiology assessment - reticulospinal tract — Kinematics and reticular spinal motor excitability
  Arms: Reaction time evaluation during non-invasive spinal cord stimulation and leg movements
Other: Training with some stimulation — Motor task combined with real or sham stimulation

SUMMARY:
Spinal cord injury leads to long-lasting paralysis and impairment. Re-enabling movement of paralyzed areas is challenging and more information is needed about neurological recovery. The purpose of this study is to understand the contribution of individual neural tracts to movements facilitated by transcutaneous spinal cord stimulation (SCS).

DETAILED DESCRIPTION:
Spinal cord injury leads to long-lasting motor impairment and paralysis that currently is not "curable". Electrical spinal cord stimulation (SCS) is beginning to be used as a neuromodulation technique to re-enable movement of paralyzed areas, however the mechanisms of neurorecovery induced by electrical neuromodulation of the spinal cord remain poorly understood. The goal of this project is to generate evidence-based knowledge of changes in the short-term excitability of corticospinal and reticulospinal neural structures that may mediate immediate improvements in motor function enabled by SCS. The proposed study will: (1) determine which kinds of SCS-facilitated movements are mediated by the corticospinal tract. (2) determine which kinds of SCS-facilitated movements are mediated by the reticulospinal tract. Having a better understanding of the neural mechanisms that are enhanced by SCS can allow the development of therapies that directly target the excitability and plasticity states of these structures towards improved and accelerated recovery.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Age between 16-65
* Healthy individuals with no major conditions of any organ system

Exclusion Criteria:

Healthy volunteers

* Not willing or able to provide consent
* Any acute or chronic pain condition
* Any acute or chronic disease of a major organ system
* Use of analgesics within 24 hours prior to study appointment
* Use of caffeine with 3 hours of study appointment
* History of epilepsy
* Implanted metal
* Active medical problems

Inclusion criteria:

Participants with spinal cord injury (SCI)

* Age between 16-65
* Traumatic SCI C4-T9 level, complete (ASIA A) or incomplete (ASIA B, C or D)
* at least 1 year post injury
* Stable medical condition
* difficulty independently performing leg movements in routine activities
* able to follow simple commands
* able to speak and respond to questions

Exclusion criteria:

Participants with spinal cord injury (SCI)

* Not willing or able to provide consent
* Any acute or chronic pain condition
* Any acute or chronic disease of a major organ system
* Use of analgesics within 24 hours prior to study appointment
* Use of caffeine with 3 hours of study appointment
* Presence of tremors, spasms and other significant involuntary movements
* Etiology of SCI other than trauma
* Concomitant neurologic disease such as traumatic brain injury (TBI) that will significantly impact the ability to follow through on study directions, multiple sclerosis (MS), stroke or peripheral neuropathy)
* History of significant medical illness (cardiovascular disease, uncontrolled diabetes, uncontrolled hypertension, osteoporosis, cancer, chronic obstructive pulmonary disease, severe asthma requiring hospitalization for treatment, renal insufficiency requiring dialysis, autonomic dysreflexia, etc).
* Severe joint contractures disabling or restricting lower limb movements.
* Unhealed fracture, contracture, pressure sore, urinary tract infection or other uncontrolled infections, other illnesses that might interfere with lower extremity exercises or testing activities
* Depression, anxiety, or cognitive impairment
* Deficit of visuo-spatial orientation
* Sitting tolerance less than 1 hour
* Severe hearing or visual deficiency
* Miss more than 3 appointments without notification
* Unable to comply with any of the procedures in the protocol
* Botulinum toxin injection in lower extremity muscles in the prior six months
* Any passive implants (osteosynthesis material, metallic plates or screws) below T9.
* Any implanted stimulator in the body (pacemaker, vagus nerve stimulator, etc.)
* History of alcoholism or another drug abuse
* Pregnancy (or possible pregnancy)
* Having an Intrathecal Baclofen Therapy Pump (ITB pump)
* History of epilepsy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Seanez, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from flyers and word of mouth at Washington University in St. Louis. The first participant was enrolled on 06/23/2022, the last participant was enrolled on 03/06/2023.
Pre-assignment Details: Recruitment was only perform for the second arm of the study: evaluating reticulospinal tract contributions during different types of movements.
  Participants performed range-of-motion and precision-control tasks in randomized order during the same session.
  As this study was terminated early based on change in funding, no participants were assigned to the "Evaluation of Motor Evoked Potentials" arm, and no data could be provided for this outcome measure.
Groups:
- Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements: This arm will receive a loud auditory stimuli to evaluate the excitability of the reticulospinal tract during non-invasive spinal cord stimulation
  Electrophysiology assessment - reticulospinal tract contribution during hip range of motion task Electrophysiology assessment - reticulospinal tract contribution during hip precision control task
  Electrophysiology assessment - reticulospinal tract contribution during plantarflexion range of motion task Electrophysiology assessment - reticulospinal tract contribution during plantarflexion precision control task
  Electrophysiology assessment - reticulospinal tract contribution during dorsiflexion range of motion task Electrophysiology assessment - reticulospinal tract contribution during dorsiflexion precision control task
- Evaluation of Motor Evoked Potentials During Non-invasive Spinal Cord Stimulation and Leg Movements: This arm will receive the transcranial magnetic stimulation to evaluate the excitability of the corticospinal tract during non-invasive spinal cord stimulation
  Electrophysiology assessment - reticulospinal tract contribution during hip range of motion task Electrophysiology assessment - reticulospinal tract contribution during hip precision control task
  Electrophysiology assessment - reticulospinal tract contribution during plantarflexion range of motion task Electrophysiology assessment - reticulospinal tract contribution during plantarflexion precision control task
  Electrophysiology assessment - reticulospinal tract contribution during dorsiflexion range of motion task Electrophysiology assessment - reticulospinal tract contribution during dorsiflexion precision control task
Period: Overall Study
Arm/Group | Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements | Evaluation of Motor Evoked Potentials During Non-invasive Spinal Cord Stimulation and Leg Movements
Started | 20 | 0
Withdrawals | 1 (One participant withdrew as they could not tolerate stimulation.) | 0
Exclusions | 3 (Three participants were excluded from the analysis: Two participants did not follow instructions, and another was excluded as an outlier based on slow reaction times across all conditions.) | 0
Completed | 19 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated early due to change in fundion. Therefore, no participants were enrolled for the evaluation of motor evoked potentials, and no data can be reported.
Groups:
- Evaluation of Motor Evoked Potentials During Non-invasive Spinal Cord Stimulation and Leg Movements: Evaluation of motor evoked potentials during non-invasive spinal cord stimulation and leg movements
  This arm will receive the transcranial magnetic stimulation to evaluate the excitability of the corticospinal tract first then the arm will receive the loud auditory stimuli to evaluate the excitability of the reticulospinal track second.
  Electrophysiology assessment - corticospinal tract: Kinematics and cortical spinal motor excitability
  Training with some stimulation: Motor task combined with real or sham stimulation
- Total: Total of all reporting groups
Arm/Group | Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements | Evaluation of Motor Evoked Potentials During Non-invasive Spinal Cord Stimulation and Leg Movements | Total
Number analyzed (Participants) | 20 | 0 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 0 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (8.67) |  | 25.8 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  | 6
  Male | 14 |  | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 |  | 2
  Not Hispanic or Latino | 18 |  | 18
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 9 |  | 9
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 11 |  | 11
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 |  | 20

OUTCOME MEASURES:

1. Primary Outcome: Changes in Corticospinal Tract Excitability After Training
Description: This primary outcome is a measure of changes in corticospinal tract excitability as quantified by changes in the amplitude size of motor evoked potentials.
  Data for this arm were not collected due to early study termination.
Time Frame: 30 minutes before and 30 minutes into intervention
Reporting Status: Not Posted

2. Primary Outcome: Reticulospinal Tract Excitability During Different Types of Movements
Description: This primary outcome measures changes in reticulospinal tract excitability (RST) during training as quantified by changes in reaction time after a startling auditory stimulus.
  RST contrubution was evaluated for dorsiflexion, plantarflexion, hip flexion movements during precision and range of motion control tasks under three conditions: with transcutaneous spinal cord stimulation or without stimulation. All conditions/evaluations were performed in the same session. 30 repetitions were performed per condition during a single session and averaged for each participant.
  RST is a ratio calculated by = (visual - startle)/(visual - auditory), where:
  visual represents the reaction time to a visual cue, auditory represents the reaction time to an auditory cue, startle represents the reaction time to a startling cue.
  A RST ratio value greater than 1 would indicate a significant contribution of the reticulospinal tract for a given task. A value equal or lower than 1 would suggest
Time Frame: During intervention, *1 Day*.
Population: The average across all participants is reported.
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements
Number analyzed (Participants) | 16
arbitrary units
  RST: Hip flexion - range of motion - No stimulation | 1.405 (0.285)
  RST: Hip flexion - precision control - No stimulation | 1.480 (0.325)
  RST: Plantar flexion - range of motion - No stimulation | 1.443 (0.325)
  RST: Plantar flexion - precision control - No stimulation | 1.455 (0.258)
  RST: Dorsiflexion - range of motion - No stimulation | 1.544 (0.578)
  RST: Dorsiflexion - precision control - No stimulation | 1.364 (0.377)
  RST: Hip flexion - range of motion - stimulation | 1.497 (0.569)
  RST: Hip flexion - precision control - stimulation | 1.689 (0.667)
  RST: Plantar flexion - range of motion - stimulation | 1.465 (0.667)
  RST: Plantar flexion - precision control - stimulation | 1.376 (0.285)
  RST: Dorsiflexion - range of motion - stimulation | 1.363 (0.225)
  RST: Dorsiflexion - precision control - stimulation | 1.294 (0.189)
Statistical Analysis 1: Comparison: Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements; Reticulospinal tract (RST) contribution computed as RST = (visual - startle)/(visual - auditory) reaction times, where a RST value greater than 1 would indicate a significant contribution of the reticulospinal tract for a given task. A one sample t-test (or Wilcoxon signed-rank test for non-normally distributed data) was used to test the hypothesis that the RST contribution for a given movement was significantly greater than 1; Test type: Superiority; p < 0.05, t-test, 2 sided — p-values have not been adjusted for multiple comparisons; Mean Difference (Final Values) = 0.405, Standard Deviation 0.285 — Difference of RST from 1 for hip range of motion task without stimulation

ADVERSE EVENTS:
Time Frame: Data were collected for single sessions (1 day) for each participant.
Description: Adverse events were monitored during each session.
Arm/Group | Reaction Time Evaluation During Non-invasive Spinal Cord Stimulation and Leg Movements | Evaluation of Motor Evoked Potentials During Non-invasive Spinal Cord Stimulation and Leg Movements
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/20 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated early due to a transition to a new grant with overlapping effort. Therefore, while some data was collected for Aim 2, no data was collected for Aim 1. The statistical analysis was not completed during the duration of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT05354206/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05354206/ICF_001.pdf